CLINICAL TRIAL: NCT00328172
Title: A Randomized, Double-blind, Placebo-controlled, Five Parallel Group Study Investigating the Efficacy and Safety of BI 1356 BS (0.5 mg, 2.5 mg and 5.0 mg Administered Orally Once Daily) Over 12 Weeks in Drug Naive and Treated Patients With Type 2 Diabetes With Insufficient Glycemic Control (Study Includes an Open-label Metformin Treatment Arm)
Brief Title: Efficacy and Safety of 3 Doses of BI1356 (Linagliptin) in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.5
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (5):
- Placebo (Placebo Comparator): Placebo tablets matching BI 1356
  Interventions: Drug: Placebo
- BI 1356 0.5 mg (Experimental): BI 1356 dose 1 once daily
  Interventions: Drug: BI 1356 dose 1 once daily
- BI 1356 2.5 mg (Experimental): BI 1356 dose 2 once daily
  Interventions: Drug: BI 1356 dose 2 once daily
- BI 1356 5.0 mg (Experimental): BI 1356 dose 3 once daily
  Interventions: Drug: BI 1356 dose 3 once daily
- Metformin (Active Comparator): Metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo — Placebo matching BI 1356
  Arms: Placebo
Drug: BI 1356 dose 3 once daily — BI 1356 dose 3 once daily
  Arms: BI 1356 5.0 mg
Drug: BI 1356 dose 2 once daily — BI 1356 dose 2 once daily
  Arms: BI 1356 2.5 mg
Drug: BI 1356 dose 1 once daily — BI 1356 dose 1 once daily
  Arms: BI 1356 0.5 mg
Drug: Metformin — Metformin
  Arms: Metformin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of several doses of BI 1356 BS (0.5, 2.5 and 5 mg daily) compared to placebo over 12 weeks of treatment in patients with Type 2 diabetes and insufficient glycemic control. In addition, there will be an open-label treatment arm with metformin for sensitivity measurement with this patient population. Population pharmacokinetics of BI 1356 BS will also be assessed in this study.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with a diagnosis of Type 2 diabetes treated only with diet and exercise (drug naïve) or with one or two oral hypoglycemic agents (as single treatment or in combination) other than rosiglitazone or pioglitazone -treatment. Antidiabetic therapy has to be stable for at least 10 weeks prior to screening.
2. Diagnosis of Type 2 diabetes with duration of at least 3 months
3. Glycosylated haemoglobin A1 (HbA1c) of:

   7.5-10.0% at screening for drug naïve patients (no wash-out needed) 7.0-9.0% at screening for patients treated with only one oral antidiabetic agent (wash-out required) 6.5-8.0% at screening for patients treated with two oral antidiabetic agents (wash-out required)
4. HbA1c of 7.5%-10.0% at Visit 3 (beginning of the 2-week placebo run-in period).
5. Age >=21 and <=75 years.
6. BMI (Body Mass Index) >=25.0 and <=40 kg/m2.
7. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Clinically relevant cardiovascular disease (e.g., myocardial infarction, stroke or transient ischemic attack within six months before enrollment)
2. Impaired hepatic function defined by serum levels of either alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase above 3-fold upper limit of normal
3. Renal insufficiency or impaired renal function defined by serum creatinine above upper limit of normal at screening
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or clinically relevant neurologic disorders (including cerebrovascular but with the exception of polyneuropathy) that would interfere with participation in the trial
5. Chronic or clinically relevant acute infections (e.g., Human immunodeficiency virus, Hepatitis)
6. History of relevant allergy/hypersensitivity that would interfere with trial participation (including allergy to investigational product or its excipients)
7. Treatment with rosiglitazone or pioglitazone within 6 months prior to screening
8. Treatment with insulin within 3 months prior to screening
9. Alcohol or drug abuse within the last 3 months that would interfere with trial participation)
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Fasting plasma glucose >240 mg/dl (= 13.3 mmol/L) at Visit 2, 3 or 4 any visit and confirmed by a second measurement (not on the same day)
12. Pre-menopausal women (last menstruation <=1 year prior to signing informed consent) who:

    1. are not surgically sterile,
    2. or are nursing or pregnant;
    3. or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra-uterine devices, oral, implantable or injectable contraceptives and vasectomised partner. No exception will be made.
13. Intolerance of metformin

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (71):
- United States (34):
  - 1218.5.10020 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.5.10001 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1218.5.10007 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1218.5.10041 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1218.5.10018 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1218.5.10016 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1218.5.10003 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.5.10011 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.5.10012 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1218.5.10017 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1218.5.10008 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 1218.5.10024 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1218.5.10039 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1218.5.10032 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1218.5.10025 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 1218.5.10034 Boehringer Ingelheim Investigational Site, Butte, Montana
  - 1218.5.10009 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1218.5.10042 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1218.5.10029 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 1218.5.10004 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1218.5.10026 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1218.5.10035 Boehringer Ingelheim Investigational Site, Mentor, Ohio
  - 1218.5.10023 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1218.5.10030 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.5.10044 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1218.5.10033 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1218.5.10038 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1218.5.10006 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.5.10040 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.5.10036 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.5.10021 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1218.5.10027 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 1218.5.10022 Boehringer Ingelheim Investigational Site, Federal Way, Washington
  - 1218.5.10014 Boehringer Ingelheim Investigational Site, Renton, Washington
- Australia (6):
  - 1218.5.61001 Boehringer Ingelheim Investigational Site, Miranda, New South Wales
  - 1218.5.61005 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1218.5.61006 Boehringer Ingelheim Investigational Site, Dandenong, Victoria
  - 1218.5.61007 Boehringer Ingelheim Investigational Site, East Ringwood, Victoria
  - 1218.5.61004 Boehringer Ingelheim Investigational Site, Fremantle, Western Australia
  - 1218.5.61002 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Canada (15):
  - 1218.5.11011 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.5.11016 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.5.11003 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1218.5.11004 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.5.11013 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.5.11015 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1218.5.11005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.5.11014 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1218.5.11010 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1218.5.11009 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.5.11012 Boehringer Ingelheim Investigational Site, Thornhill, Ontario
  - 1218.5.11002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.5.11006 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1218.5.11017 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
  - 1218.5.11018 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Czechia (5):
  - 1218.5.42002 Boehringer Ingelheim Investigational Site, Olomouc
  - 1218.5.42003 Boehringer Ingelheim Investigational Site, Prague
  - 1218.5.42004 Boehringer Ingelheim Investigational Site, Prague
  - 1218.5.42005 Boehringer Ingelheim Investigational Site, Prague
  - 1218.5.42001 Boehringer Ingelheim Investigational Site, Sternberk
- Russia (5):
  - 1218.5.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.5.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.5.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.5.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.5.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Ukraine (6):
  - 1218.5.38005 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.5.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.5.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.5.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.5.38004 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.5.38006 Boehringer Ingelheim Investigational Site, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin (BI 1356) 0.5 mg: Patients randomized to receive treatment with linagliptin 0.5 mg
- Linagliptin (BI 1356) 2.5 mg: Patients randomized to receive treatment with linagliptin 2.5 mg
- Linagliptin (BI 1356) 5.0 mg: Patients randomized to receive treatment with linagliptin 5.0 mg
- Metformin: Patients randomized to receive treatment with metformin
Period: Overall Study
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin
Started | 67 | 58 | 57 | 55 | 65
Completed | 45 | 44 | 47 | 42 | 60
Not Completed | 22 | 14 | 10 | 13 | 5
Not completed — Adverse Event | 3 | 2 | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 6 | 0
Not completed — Lack of Efficacy | 14 | 9 | 4 | 4 | 3
Not completed — Other reason (not specified) | 3 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin | Total
Number analyzed (Participants) | 67 | 58 | 57 | 55 | 65 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (8.9) | 58.0 (9.4) | 59.8 (10.3) | 56.6 (9.6) | 53.7 (10.7) | 57.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 13 | 30 | 24 | 26 | 127
  Male | 33 | 45 | 27 | 31 | 39 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic | 63 | 54 | 51 | 49 | 61 | 278
  Hispanic | 4 | 4 | 6 | 6 | 4 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 52 | 53 | 52 | 57 | 272
  Black | 6 | 3 | 3 | 1 | 5 | 18
  Asian | 3 | 3 | 1 | 2 | 2 | 11
  Missing | 0 | 0 | 0 | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/square meter] | 30.8 (4.1) | 30.9 (3.8) | 31.5 (4.5) | 31.2 (4.3) | 31.2 (4.8) | 31.1 (4.3)
Baseline glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] | 8.3 (0.63) | 8.2 (0.62) | 8.4 (0.80) | 8.4 (0.80) | 8.3 (0.64) | 8.3 (0.69)
Fasting blood plasma glucose (FPG) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] | 183.0 (34.9) | 185.2 (34.0) | 191.9 (37.8) | 188.7 (40.1) | 193.9 (45.9) | 188.4 (38.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) at Week 12
Description: The change from baseline reflects the Week 12 HbA1c minus the Week 0 HbA1c. Means are adjusted for baseline HbA1c.
Time Frame: Baseline, week 12
Population: Full Analysis Set includes all randomized patients with baseline and on-treatment value of HbA1c. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin
Number analyzed (Participants) | 63 | 57 | 55 | 54 | 65
percent | 0.18 (0.10) | 0.04 (0.10) | -0.24 (0.10) | -0.28 (0.10) | -0.68 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356) 0.5 mg; Linagliptin 0.5 mg versus placebo; Test type: Superiority or Other; p = 0.3271, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline HbA1c as a linear covariate; Mean Difference (Final Values) = -0.14, 95% CI [-0.41 to 0.14]
Statistical Analysis 2: Comparison: Placebo vs Linagliptin (BI 1356) 2.5 mg; Linagliptin 2.5 mg versus placebo; Test type: Superiority or Other; p = 0.0032, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline HbA1c as a linear covariate; Mean Difference (Final Values) = -0.42, 95% CI [-0.69 to -0.14]
Statistical Analysis 3: Comparison: Placebo vs Linagliptin (BI 1356) 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0012, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline HbA1c as a linear covariate; Mean Difference (Final Values) = -0.46, 95% CI [-0.74 to -0.18]
Statistical Analysis 4: Comparison: Placebo vs Metformin; Metformin versus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline HbA1c as a linear covariate; Mean Difference (Final Values) = -0.85, 95% CI [-1.1 to -0.59]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: Change from baseline reflects the Week 12 FPG minus the Week 0 FPG. Means are adjusted for baseline FPG.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin
Number analyzed (Participants) | 63 | 57 | 55 | 54 | 65
mg/dL | 4.24 (4.4) | 6.69 (4.6) | -15.2 (4.7) | -9.09 (4.8) | -30.1 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356) 0.5 mg; Linagliptin 0.5 mg versus placebo; Test type: Superiority or Other; p = 0.7027, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline FPG as a linear covariate; Mean Difference (Final Values) = 2.45, 95% CI [-10 to 15.1]
Statistical Analysis 2: Comparison: Placebo vs Linagliptin (BI 1356) 2.5 mg; Linagliptin 2.5 mg versus placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline FPG as a linear covariate; Mean Difference (Final Values) = -19.4, 95% CI [-32 to -6.6]
Statistical Analysis 3: Comparison: Placebo vs Linagliptin (BI 1356) 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0418, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline FPG as a linear covariate; Mean Difference (Final Values) = -13.3, 95% CI [-26 to -0.5]
Statistical Analysis 4: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model includes treatment as a fixed classification effect and baseline FPG as a linear covariate; Mean Difference (Final Values) = -34.3, 95% CI [-47 to -22]

3. Secondary Outcome: Percentage of Patients With Absolute Efficacy Response (HbA1c <= 7.0%) at 12 Weeks
Description: An absolute efficacy response is defined as HbA1c <= 7.0% at 12 weeks. A non-response is defined as HbA1c > 7.0% at 12 weeks.
Time Frame: Baseline, week 12
Population: FAS patients with baseline HbA1c > 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: participants
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin
Number analyzed (Participants) | 63 | 57 | 55 | 54 | 65
participants
  HbA1c <= 7% | 6.3 | 10.5 | 7.3 | 11.1 | 26.2
  HbA1c > 7% | 93.7 | 89.5 | 92.7 | 88.9 | 73.8
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356) 0.5 mg; Linagliptin 0.5 mg versus placebo; Test type: Superiority or Other; p = 0.413, Regression, Logistic; Odds Ratio (OR) = 1.735, 95% CI [0.464 to 6.492]
Statistical Analysis 2: Comparison: Placebo vs Linagliptin (BI 1356) 2.5 mg; Linagliptin 2.5 mg versus placebo; Test type: Superiority or Other; p = 0.842, Regression, Logistic; Odds Ratio (OR) = 1.157, 95% CI [0.275 to 4.861]
Statistical Analysis 3: Comparison: Placebo vs Linagliptin (BI 1356) 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.364, Regression, Logistic; Odds Ratio (OR) = 1.844, 95% CI [0.492 to 6.910]
Statistical Analysis 4: Comparison: Placebo vs Metformin; Metformin versus placebo; Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 5.224, 95% CI [1.648 to 16.562]

ADVERSE EVENTS:
Time Frame: First dose of study medication up to a period of 30 days after the last dose of study medication, an average of 106 days
Arm/Group | Placebo | Linagliptin (BI 1356) 0.5 mg | Linagliptin (BI 1356) 2.5 mg | Linagliptin (BI 1356) 5.0 mg | Metformin
Serious Adverse Events (participants affected / at risk) | 1/67 | 1/58 | 2/57 | 0/55 | 1/65
Other Adverse Events (participants affected / at risk) | 18/67 | 15/58 | 9/57 | 8/55 | 13/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Linagliptin (BI 1356) 0.5 mg (N=58) | Linagliptin (BI 1356) 2.5 mg (N=57) | Linagliptin (BI 1356) 5.0 mg (N=55) | Metformin (N=65)
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Linagliptin (BI 1356) 0.5 mg (N=58) | Linagliptin (BI 1356) 2.5 mg (N=57) | Linagliptin (BI 1356) 5.0 mg (N=55) | Metformin (N=65)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 5
Influenza (Infections and infestations) | 1 | 1 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 1 | 0
Blood glucose increased (Investigations) | 4 | 2 | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 7 | 2 | 1 | 3
Headache (Nervous system disorders) | 1 | 5 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.